CLINICAL TRIAL: NCT05938946
Title: A Phase I, Randomized, Double-blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of L608 for Inhalation in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of L608 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmosa Biopharm Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PBI L608p1
Record Dates: First submitted 2023-06-09; First posted 2023-07-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, double-blinded, single ascending dose escalation
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded, single ascending dose escalation design. After confirmation of eligibility, subjects will be randomized at a ratio of 1:1 (for sentinel dosing) followed by 5:1 for rest of the cohorts to receive the assigned dose of L608 or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L608 Liposomal inhalation solution (Experimental): Eight subjects will be enrolled in each cohort and be randomized to receive assigned dose of L608 or placebo (6:2).
  Interventions: Drug: L608 Inhalation Solution
- Placebo (Experimental): Eight subjects will be enrolled in each cohort and be randomized to receive assigned dose of L608 or placebo (6:2).
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: L608 Inhalation Solution — subjects will be randomized at a ratio of 1:1 (for Sentinel dosing) followed by 5:1 for rest of the cohort to receive the assigned dose of L608 or placebo
  Arms: L608 Liposomal inhalation solution
Drug: Placebo solution — subjects will be randomized at a ratio of 1:1 (for Sentinel dosing) followed by 5:1 for rest of the cohort to receive the assigned dose of L608 or placebo
  Arms: Placebo

SUMMARY:
This is a Phase I, randomized, double-blinded, placebo-controlled single ascending dose, sequential-group study to evaluate the safety, tolerability, and PK of single ascending doses of L608 inhalation in healthy volunteers.

DETAILED DESCRIPTION:
L608 inhalation Solution (L608) is developed by Pharmosa Biopharm Inc. (PBI) as a new liposomal Iloprost formulation for inhalation use in the treatment of patients with PAH (WHO Group 1). As a liposomal formulation of iloprost, L608 is intended to reduce the dosing frequency, as well as provide sustained and selective release along with achieving therapeutically relevant iloprost level. Meanwhile, L608 is expected to mitigate burst release related local irritation and systemic side effects (e.g., hypotension due to plasma peak) in clinical practice.

This Phase I, randomized, double-blinded, placebo-controlled study will be conducted in healthy volunteers in Australia to evaluate the safety, tolerability, and pharmacokinetic of L608. The dose escalation design is applied in this study. The sentinel dosing design will be applied for all cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women aged between 18 and 65 (inclusive) at the time of Screening visit. Females must not be pregnant or lactating.
2. Body Mass Index (BMI) of ≥18.5 and ≤30.0 kg/m2
3. Non-smokers or former smokers who have smoked ≤ 100 cigarettes in their lifetime and have not consumed any tobacco or tobacco-containing products for at least 3 months prior to Screening.
4. Females must not be pregnant or lactating and must use acceptable, highly effective double contraception from Screening until 3 months after the last dose of the Investigational product.

Key Exclusion Criteria:

1. Subjects with contraindications or sensitivity to any components of the study treatment.
2. Subjects with medical histories (within 3 months prior to Screening) or ongoing conditions of any clinically significant and/or any other medical conditions which may jeopardize the safety of the subjects and/or effect the results of the study at the Investigator's discretion.
3. Subjects with histories or active conditions of unexplained bleeding events, hemoptysis, abnormal bleeding tendencies, and/or coagulation disorders.
4. Subjects who voluntarily participate in this study and sign the informed consent form prior to any study procedures.
5. Subjects with histories or active conditions of asthma, sleep apnea, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, bronchiectasis, bronchospasm, and/or reactive airway. Subjects who have had childhood asthma which have resolved as deemed by the PI can be considered.
6. Subjects with histories or active conditions of myocardial infarction (MI), cerebrovascular accident (CVA), coronary artery disease (CAD), unstable angina, heart failure, significant cardiac arrhythmias, congenital or acquired valvular heart disease with clinically insignificant symptom, suspected lung congestion, and/or pulmonary arterial hypertension (PAH) causing by venous thromboembolism.
7. Subjects with systolic blood pressure < 90 mmHg or > 160 mmHg and/or diastolic blood pressure < 50 mmHg or > 95 mmHg at Screening or check-in visit.
8. Subjects with FEV1 less than 80% predicted, FVC ˂80% predicted, or resting oxygen saturation less than 95% at Screening or check-in visit.
9. Subjects with histories of drug or alcohol abuse within 1 year prior to subject check-in (Day -1). Regular alcohol consumption defined as > 10 standard drinks per week.
10. Consumption of products containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing and products containing grapefruit and/or pomelo (shown to inhibit cytochrome P450 [CYP] 3A4 activity) within 10 days prior to drug administration.
11. Positive results of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), and pregnancy test.
12. Blood donation or significant blood loss (>480 ml) within 3 months prior to Screening.
13. Subjects are pregnant or breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicity (DLT) | Baseline to Day 14
  The percentage of subjects with dose limiting toxicity (DLT) within 14 days after dosing
The incidence of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline to Day 21
  The percentage of subjects with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) within 21 days after dosing.
Frequency and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Baseline to Day 21
  The frequency and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) within 21 days after dosing.

SECONDARY OUTCOMES:
AUC0-t | Baseline to 24 hours
  Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration
AUC0-∞ | Baseline to 24 hours
  Area under the plasma concentration-time curve from time 0 to infinity
%AUCextrap | Baseline to 24 hours
  AUC extrapolated from the last measurable concentration to infinity as a percentage of total AUC
Cmax | Baseline to 24 hours
  Maximum observed plasma concentration
Tmax | Baseline to 24 hours
  Time to reach the maximum observed plasma concentration
T1/2 | Baseline to 24 hours
  Apparent plasma terminal elimination half-life
CL/F | Baseline to 24 hours
  Apparent total plasma clearance
Vz/F | Baseline to 24 hours
  Apparent volume of distribution during the terminal phase
kel | Baseline to 24 hours
  Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia